CLINICAL TRIAL: NCT00124618
Title: Cetuximab (C225) and Radiation in Elderly and /or Poor Performance Status Patients With Locally Advanced Non-Small Cell Lung Cancer: A Phase II Study to Evaluate Survival and Toxicity
Brief Title: Cetuximab and Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0422; NCI-2012-02664 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000435991 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab/Radiation (Experimental): Cetuximab (C225) and Radiation
  Interventions: Biological: cetuximab; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cetuximab together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with radiation therapy works in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 11 month survival rate in older and/or poor performance status patients with stage IIIA or stage IIIB non-small cell lung cancer treated with cetuximab and radiotherapy.

Secondary

* Determine the tumor response rate, overall survival, and time to disease progression in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine whether fear of death is less severe in the oldest of patients treated with this regimen.
* Determine whether fear of death predicts survival of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, and 43. Beginning on day 8, patients receive concurrent radiotherapy once daily on days 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed within 1 week, at 1 and 4 months, and then every 3 months for up to 3 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 20 months

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIA or IIIB disease
* Must be a candidate for curative radiotherapy
* Not a candidate for other concurrent chemotherapy and radiotherapy
* No surgical treatment available
* No pleural effusion suspected or proven to be malignant
* No stage IV disease by bone scan or positron emission tomography scan, CT scan or MRI of the brain, and CT scan of the chest within the past 30 days

PATIENT CHARACTERISTICS:

Age * 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2 (age ≥ 65 years)
* ECOG 2 (age 18 to 64 years)

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST ≤ 3 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Pulmonary

* FEV_1 ≥ 1 L
* No idiopathic pulmonary fibrosis

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Magnesium normal
* No uncontrolled infection
* No other severe underlying disease that would preclude study entry
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or noninvasive carcinoma
* No major psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy for NSCLC

Endocrine therapy

* Not specified

Radiotherapy

* No prior therapeutic radiotherapy to the chest
* No concurrent intensity modulated radiotherapy

Other

* No prior epidermal growth factor receptor inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-01; Primary Completion 2008-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (175):
- United States (175):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Jatoi A, Schild SE, Foster N, Henning GT, Dornfeld KJ, Flynn PJ, Fitch TR, Dakhil SR, Rowland KM, Stella PJ, Soori GS, Adjei AA. A phase II study of cetuximab and radiation in elderly and/or poor performance status patients with locally advanced non-small-cell lung cancer (N0422). Ann Oncol. 2010 Oct;21(10):2040-2044. doi: 10.1093/annonc/mdq075. Epub 2010 Jun 21. PMID 20570832

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled a total of 58 patients. All patients received study treatment, and one patient was deemed ineligible during an North Central Cancer Treatment Group (NCCTG) audit. This analysis includes all 58 patients, with the exception of Overall Survival (OS), Time to Progression (TTP), and response which remove the ineligible patient.
Groups:
- Cetuximab/Radiation: Cetuximab (C225) and Radiation therapy
Period: Overall Study
Arm/Group | Cetuximab/Radiation
Started | 58
Completed | 57
Not Completed | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab/Radiation
Number analyzed (Participants) | 58
Age, Customized [Median (Full Range); unit: years]
  Median Age in years (Range) | 77 [60 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: 11-month Survival Rate
Description: Eleven-month survival was chosen as the survival endpoint in this trial because it represents an improvement over the median survival that is observed with radiation alone. 11-month survival will be considered synonymous with "success", unless specified otherwise. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. All evaluable patients will be followed from the time of protocol enrollment until death or a minimum of 11 months.
Time Frame: From baseline to 11 months.
Population: This study enrolled a total of 58 patients. All patients received study treatment, and one patient was deemed ineligible during an NCCTG audit. This analysis includes all 57 patients. Forty of 57 patients (70%) reached the 11-month survival primary point.
Measure: Number; unit: percentage of participants
Arm/Group | Cetuximab/Radiation
Number analyzed (Participants) | 57
percentage of participants | 70

2. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From baseline to up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab/Radiation
Number analyzed (Participants) | 57
months | 15.1 [13.1 to 19.3]

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death.
Time Frame: From Baseline to up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab/Radiation
Number analyzed (Participants) | 57
months | 7.2 [5.8 to 8.6]

4. Secondary Outcome: Tumor Response (Complete and Partial)
Description: A confirmed tumor response is defined to be a Complete Response (CR) or Partial Response (PR) noted as the objective status on 2 consecutive evaluations at least 3 months apart. All patients meeting the eligibility criteria who have signed a consent form and have begun treatment will be evaluable for response.
Time Frame: Baseline, 1 month and 4 months after completion of treatment and then every 3 months until Progressive Disease (PD) or up to a maximum of 3 years from registration
Measure: Number; unit: participants
Arm/Group | Cetuximab/Radiation
Number analyzed (Participants) | 57
participants
  Number of patients with Partial Response (PR) | 15
  Number of patients with Complete Response (CR) | 0

ADVERSE EVENTS:
Arm/Group | Cetuximab/Radiation
Serious Adverse Events (participants affected / at risk) | 3/58
Other Adverse Events (participants affected / at risk) | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab/Radiation (N=58)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab/Radiation (N=58)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (4)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (2)
Extraocular muscle paresis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (18)
Diarrhea (Gastrointestinal disorders) | 11 (30)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 10 (19)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 19 (47)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 3 (4)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 18 (46)
Nausea (Gastrointestinal disorders) | 25 (72)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 19 (31)
Chills (General disorders) | 2 (4)
Death NOS (General disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
Fatigue (General disorders) | 24 (68)
Pain (General disorders) | 2 (7)
Hypersensitivity (Immune system disorders) | 4 (5)
Nail infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 12 (17)
Skin infection (Infections and infestations) | 1 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 12 (24)
Lymphocyte count decreased (Investigations) | 5 (11)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 5 (16)
Weight loss (Investigations) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 13 (48)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 7 (9)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 22 (64)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (6)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (3)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (19)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 8 (15)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 18 (56)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 12 (38)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 50 (258)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (5)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes